CLINICAL TRIAL: NCT05866445
Title: An Updated Wearable Magnetic Flux Device to Optimize Blood Pressure Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart Centre Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021/2396
Record Dates: First submitted 2023-05-10; First posted 2023-05-19 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2024-11

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Participants from 2 different groups (Hypertensive and Normotensive groups) will be randomized into 2:1:1 to receive the original strength magnetic device vs half strength magnetic device (half the strength of the original magnetic device) vs the sham device respectively.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Study team and participants will be blinded to whether they are receiving the magnetic device or sham device. Delegated unblinded team member will assign study device to recruited participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hypertensive (Experimental): Hypertensive patients
  Interventions: Device: Wearable BP device; Device: 24-hour ambulatory blood pressure monitor
- Normotensive participants (Experimental): Normotensive participants with no high blood pressure
  Interventions: Device: Wearable BP device; Device: 24-hour ambulatory blood pressure monitor

INTERVENTIONS:
Device: Wearable BP device — Wearable study BP device to be worn for 8 hours within study participation.
Device: 24-hour ambulatory blood pressure monitor — 24-hour ambulatory blood pressure monitor to be worn for 24-hours during study participation.

SUMMARY:
The goal of this study involving a wearable magnetic flux device is to study the impact of static magnetic flux on blood pressure control in hypertensive and normotensive populations. The main objectives are:

1. Study the safety and efficacy of static magnetic flux on blood pressure control in normal and hypertensive patients.
2. Incorporate this into a portable, wearable device to increase availability and outreach.

Participants will be required to wear a wearable BP device, an ambulatory BP and answer a questionnaire for this study. Researchers will compare between hypertensive and normotensive groups to achieve objective of this study.

DETAILED DESCRIPTION:
Hypertension is significant public health problem locally as well as internationally. Untreated hypertension results in much morbidity and mortality. In Singapore, there is a significant proportion of poorly controlled hypertensives, with its attendant risks. The compliance to antihypertensive medications has been reported at about only 50%. Several pertinent factors have been brought up including dislike of oral medications, having too many medications, cost of chronic medications and side effects of medications. Several studies have also pointed out the importance of combining various components (e.g. regimen simplification, patient behavioural modification, communication and education by health professionals) in order to improve antihypertensives adherence.

This project aims to study the impact of static magnetic flux on blood pressure control. If efficacious, this may potentially provide an effective, non-invasive, non-pharmacological option for blood pressure control. In addition, the project aims to incorporate this static magnetic flux into a wearable, portable device to increase its availability and uptake. This may potentially increase compliance amongst patients who may be non-compliant to oral medications, and help reduce the attendant mortality and morbidity associated with hypertension.

In this double-blind randomized control trial, 200 participants (140 hypertensive, 60 normotensive) will be recruited. Participants will be randomized into 2:1:1 to receive the original strength magnetic device vs half strength magnetic device (half the strength of the original magnetic device) vs the sham device respectively. The half strength arm will allow us to evaluate the dose-response effect of the magnetic field. The magnetic and sham devices will be made identical in appearance and numbered for assignment purposes during the period of the trial. Study team and participants will be blinded to whether they are receiving the magnetic device or sham device.

The study participation will consist of 2 visits, an initial visit and device return visit. The participants will wear a 24hr ambulatory blood pressure (ABP) monitor for 24 hours, whereas the study device will be worn only for 8 hours. Prior to that, a blood pressure measurement will be taken at rest to confirm eligibility. Baseline ABP measurement will be taken for 3-4 hours, followed by the additional study device to be worn for the next 8 hours. Subsequently, participants will remove the study device leaving only the ABP monitor for the rest of the remaining hours. The first 3-4 hours will give an indication of the subject's baseline blood pressure. The next 8hr will give an indication of the effect of the device. The remainder 12-13hr will allow us to see the impact on blood pressure after the device is removed. The subjects will be required to complete a hardcopy questionnaire on their baseline demographics, characteristics, experience with the device, and any side effects.

ELIGIBILITY:
Inclusion Criteria:

* For normotensive patients, Systolic Blood Pressure 100-139mmHg/ Diastolic Blood Pressure 50-89mmHg
* For hypertensive patients, SBP 140-180mmHg, DBP 90-110mmHg (no change in blood pressure medications in last one month) OR Hypertensive patients with stable blood pressure (SBP not <100, DBP not <50) well controlled on medication

Exclusion Criteria

* SBP <100mmHg, DBP<50mmHg
* SBP>180mmHg, DBP >110mmHg
* Recent change (<1month) in blood pressure medications
* Prior stroke
* Prior ischemic heart disease
* Prior peripheral vascular heart disease
* Prior carotid stenosis or bruit
* Presence of metallic implants (e.g. ICD, pacemaker, etc)
* Pregnancy
* Breast feeding
* Allergy to device material/skin allergy

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Change of blood pressure measurement after wearing study BP device | 24 hours
  The investigators will be assessing the 24Hours ambulatory blood pressure monitor report with hourly averages to determine the outcome. Blood pressure measurements will reflect whether the wearable BP device has any impact on the participants' blood pressure before, during and after the participants wear the device.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Sheng Foo, M.D., Principal Investigator — National Heart Centre Singapore
Locations (1):
- National Heart Centre Singapore, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No